CLINICAL TRIAL: NCT04375059
Title: Therapeutic Effects of Interactive Attention Training on Children With Attention Deficit Hyperactivity Disorder
Brief Title: Effects of Attention Training on Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Principle investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019SKHADR038
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: attention training; children; therapeutic effects; developmental delay
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Learning Disabilities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): 3 months of interactive attention training programs, 2 times per week, 15 min per session, a total of 24 sessions, with conventional rehabilitation programs
  Interventions: Other: using interactive attention training system
- Control group (No Intervention): 3 months of conventional rehabilitation programs without interactive attention training programs

INTERVENTIONS:
Other: using interactive attention training system — using the interactive attention training system to children with Attention Deficit Hyperactivity Disorder
  Arms: Study group

SUMMARY:
Using a double-blind, randomized controlled design to investigate the therapeutic effects of interactive attention training for children with Attention Deficit Hyperactivity Disorder who are receiving conventional rehabilitation programs due to developmental delay.

DETAILED DESCRIPTION:
A total of 30 children with Attention Deficit Hyperactivity Disorder conducting conventional rehabilitation programs well be enrolled.

The children are randomized into two groups, including study group with conventional rehabilitation programs and interactive attention training: 2 times per week, 15 min per session, with a total of 24 sessions in 3 months; and control group with conventional rehabilitation programs without interactive attention training.

Therapeutic effects, including working memory, attention, functional performance, physical function, health-related quality of life will be evaluated at baseline, and 3 months and 6 months after the intervention.

The evaluator and children will be blinded to the group's allocation during the whole course of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* children with a diagnosis of Attention Deficit Hyperactivity Disorder with developmental delay, under regular conventional rehabilitation programs, Intelligence quotient 70 or greater

Exclusion Criteria:

* age less than 4 or greater than 8 of children diagnosed with Attention Deficit Hyperactivity Disorder with developmental delay, under regular conventional rehabilitation programs, Intelligence quotient less than 70

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of symptoms of attention deficit hyperactivity disorder | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a better outcome
  score assessed by Swanson, Nolan and Pelham questionnaire

SECONDARY OUTCOMES:
changes of sensory integration | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Sensory Profile
changes of visual motor integration | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Beery-Buktenica Visual Motor Integration Test
changes of intelligence | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Wechsler Intelligence Scale for Children
changes of functional performance | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Pediatric Outcome Data Collection Instrument
changes of health-related quality of life | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a worse outcome
  score assessed by Pediatric Quality of Life Inventory
changes of family impact | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a worse outcome
  Child Health Questionnaire, parent form 28
changes of walking speed | time change from baseline to 3 months of treatment, and 3 months after treatment
  walking speed
changes of chair climbing speed | time change from baseline to 3 months of treatment, and 3 months after treatment
  stairs climbing speed
changes of balance | time change from baseline to 3 months of treatment, and 3 months after treatment
  one leg standing time
changes of coordination | score change from baseline to 3 months of treatment, and 3 months after treatment, lower scores mean a worse outcome
  Berg Balance Scale
changes of balance and coordination | time change from baseline to 3 months of treatment, and 3 months after treatment
  timed up and go test
changes of physical performance | time change from baseline to 3 months of treatment, and 3 months after treatment
  5 time sit to stand test

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Ru-Lan, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No